CLINICAL TRIAL: NCT05373043
Title: Evaluating the Long-term Health Consequences of COVID-19 and Rehabilitation Therapies to Speed Convalescence
Brief Title: Long-term COVID and Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F3810-R; RX003810 (Other Grant/Funding Number: Veteran Affairs)
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Long-COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Aim 1: Participants will be either long-COVID (n=40), COVID recovered (n=40), or Controls who never had COVID (n=40) and testing will take place at baseline, months 3 and 6, and every 6 months thereafter until the end of year 4. Peripheral and cerebral vascular endothelial function, along with neurocognitive testing, pulmonary function, physical function, and quality of life, will be assessed at baseline, months 3 and 6, and then every 6 months for four years.
  Aim 2: Participants will be either long-COVID (n=60), COVID-recovered (n=60), or Controls who avoided COVID (n=60) as defined in Aim 1. Participants will be assigned to the Exercise+Placebo or Exercise+Mito-Q rehabilitation interventions using block randomization (block size 10). This will provide equal sample sizes (n=30) per intervention for each group.
Who Masked: Participant, Investigator
Masking Description: Aim 2 will be a double blind placebo controlled design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Rehabilitation (Experimental): Participants will be assigned to the Exercise+Placebo or Exercise+Mito-Q rehabilitation interventions using block randomization (block size 10).
  Interventions: Dietary Supplement: Mitoquinone
- Exercise Rehabilitation with Placebo (Placebo Comparator): Participants will be assigned to Exercise+Placebo rehabilitation using block randomization (block size 10)
  Interventions: Dietary Supplement: Mitoquinone; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitoquinone — Mito-Q is a supplement that targets mitochondrial function. Linking a triphenyl-phosphonium cation to coenzyme-Q, to produce Mito-Q, results in a lipophilic compound, which, due to the large mitochondrial membrane potential, selectively accumulates within mitochondria. This targeted antioxidant approach results in 50- to 100-fold more Mito-Q accumulation compared to non-targeted antioxidant delivery.
  Other Names: MitoQ
Dietary Supplement: Placebo — A placebo will be used in combination with exercise rehabilitation allowing for a double blinded placebo controlled design.
  Arms: Exercise Rehabilitation with Placebo

SUMMARY:
The proposed focuses on improving both morbidity and mortality in older Veterans and those recovering from COVID-19 by developing rehabilitation therapies to augment vascular endothelial function by combating the oxidative stress and inflammation associated with aging and further induced by COVID-19. The investigators expected outcomes will have an important positive impact because they will provide scientifically sound recommendations for rehabilitation to improve vascular endothelial function and minimize the long-term consequences of COVID-19.

DETAILED DESCRIPTION:
COVID-19 induces profound vascular endothelial dysfunction, the long-term impact of which is unknown.

Moreover, recovery from COVID-19 is delayed in a substantial number of COVID-19 patients (~ 30-40%) and characterized by persistent symptoms of fatigue, weakness, and neurocognitive deficits commonly referred to as "long-COVID". The overall objective of this project is to evaluate the long-term consequences of COVID-19 in older Veterans and provide scientifically sound recommendations for vascular endothelial function-based rehabilitation in older Veterans after COVID-19 and older Veterans in general. The central hypothesis is that, given the fundamental role of oxidative stress and inflammation in long-COVID, vascular endothelial dysfunction following COVID-19 will be associated with long-term negative impacts on health and exercise-based rehabilitation with mitochondria-targeted antioxidant (Mito-Q) supplementation will synergistically improve peripheral and cerebral vascular endothelial dysfunction in older Veterans while convalescing from COVID-19. The rationale for this project is that improving COVID-19-induced vascular endothelial dysfunction by decreasing oxidative stress and inflammation with optimized rehabilitation has the potential to improve health in Veterans with long-COVID, and improve both morbidity and mortality in older Veterans. The central hypothesis will be tested by pursuing two Specific Aims: 1) determine the time course and health risks of vascular endothelial dysfunction in older Veterans with long-COVID, older Veterans who are COVID-recovered, and older Veterans who never had COVID and 2) determine the efficacy of exercise-based rehabilitation with and without Mito-Q supplementation to improve vascular endothelial function in older Veterans with long-COVID, older Veterans who are COVID-recovered, and older Veterans who never had COVID. Under Specific Aim 1, single passive leg movement (sPLM), flow-mediated dilation (FMD), and the breath-hold acceleration index (BHAI) will be used to evaluate microvascular, conduit artery, and cerebral vascular endothelial function in older patients twice annually for 4 years to determine long-term impact of COVID-19 on vascular endothelial function. Additionally, patient health risks, negative outcomes, [neurocognitive function, and pulmonary function] will be tracked during this time to determine the prognostic ability of the peripheral and cerebral vascular endothelial function assessments. For Specific Aim 2, microvascular (sPLM), conduit artery (FMD), and cerebral (BHAI) vascular endothelial function will be assessed before and after either exercise-based rehabilitation or exercise-based rehabilitation combined with Mito-Q supplementation to determine their efficacy to improve peripheral and cerebral vascular endothelial function in COVID-impacted Veterans and older Veterans in general. The research proposed in this application is innovative because it focuses on lead therapeutic candidates to rehabilitate peripheral and cerebral vascular endothelial function by combatting the underlying issue of a sustained elevation in oxidative stress and inflammation associated with aging and further impacted by COVID-19. The proposed research is significant because it is expected to provide scientifically sound recommendations for rehabilitation to improve health in older Veterans and those struggling to recover from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or greater
* Long-COVID and COVID-recovered patients must have SARS-CoV-19 positive test near the time of COVID-19 diagnosis
* Long-COVID and COVID-recovered patients must be 3-12 months post-initial COVID-19 diagnosis
* Ability to sign informed consent

Exclusion Criteria:

* BMI >45 kg/m2
* Unstable (<6 months) or severe coronary artery disease (CAD-RADS score = 4A), peripheral artery disease (Ankle Brachial Index <0.40), cerebrovascular disease (identified by previous stroke in last 12 months), severe COPD (=Stage III), uncontrolled hypertension (>160/100 mmHg), chronic kidney disease requiring dialysis, severe renal insufficiency (creatinine clearance <30 by the Cockcroft-Gault formula), Alzheimer's disease, dementia
* Orthopedic limitations that would prohibit exercise
* [Current smokers and individuals that stopped smoking in the last 10 years]
* Already taking Mito-Q or unwilling to cease dietary supplements for participation
* Any other condition or event considered exclusionary by the PIs or a physician

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Flow Mediated Dilation (FMD) | Baseline, months 3 and 6, and every 6 months thereafter until the end of year 4.
  FMD will be quantified as the peak diameter measured post-cuff release and expressed as a percent change from the baseline diameter. Higher FMD indicates better vascular function and greater change over time suggests improvement.
Change in Microvascular Function with passive leg movement (PLM) | Baseline, months 3 and 6, and every 6 months thereafter until the end of year 4.
  The PLM leg blood flow response will be characterized by the area under the curve over 45 seconds, accounting for baseline. Higher PLM indicates better vascular function and greater change over time suggests improvement.
Change in Cerebral Vascular Endothelial Function with Breath Hold Acceleration Index (BHAI) | Baseline, months 3 and 6, and every 6 months thereafter until the end of year 4.
  BHAI will be determined by fitting a linear regression to the most linear portion of the change in middle cerebral artery blood velocity over time during the breath-hold maneuver. Higher BHAI indicates better vascular function and greater change over time suggests improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Douglas Trinity, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No